CLINICAL TRIAL: NCT06332534
Title: A Phase 3 Multicenter Study to Evaluate Efficacy, Safety, and Pharmacokinetics of Upadacitinib With Open-Label Induction, Randomized, Double-Blind Maintenance and Open-Label Long-Term Extension in Pediatric Subjects With Moderately to Severely Active Crohn's Disease and Inadequate Response, Intolerance, or Medical Contraindications to Corticosteroids, Immunosuppressants, and/or Biologic Therapy
Brief Title: Crohn's Disease: Efficacy, Safety, and Pharmacokinetics of Upadacitinib in Pediatric Subjects With Moderately to Severely Active Crohn's Disease
Acronym: U-EMPOWER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-671
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Upadacitinib; RINVOQ
MeSH Terms: conditions — Crohn Disease | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Period 1: Open Label Induction Phase (Dose A) (Experimental): All participants in the open label induction phase of Period 1 will receive upadacitinib Dose A for 12 weeks based on body weight.
  Interventions: Drug: Upadacitinib
- Period 1: Double-Blind Maintenance Phase (Dose B) (Experimental): Clinical responders per PCDAI at the end of open label induction phase of Period 1 will be randomly assigned to receive Dose B or C for 52 weeks (oral solution dose will be based on body weight)
  Interventions: Drug: Upadacitinib
- Period 1: Double-Blind Maintenance Phase (Dose C) (Experimental): Clinical responders per PCDAI at the end of open label induction phase of Period 1 will be randomly assigned to receive either upadacitinib Dose C or B for 52 weeks (oral solution dose will be based on body weight)
  Interventions: Drug: Upadacitinib
- Period 2: Open Label Long-Term Extension Phase Cohort 1 (Experimental): Participants receiving double-blind maintenance therapy with upadacitinib Dose B or upadacitinib Dose C daily in Period 1 who complete the Week 64 visit will receive upadacitinib Dose B daily for up to 156 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Open Label Long-Term Extension Phase Cohort 2 (Experimental): Participants who were receiving rescue therapy with open-label upadacitinib Dose C during maintenance phase in Period 1 and completed the Week 64 visit will continue to receive upadacitinib Dose C daily for up to 156 weeks.
  Interventions: Drug: Upadacitinib
- Period 2: Open Label Long-Term Extension Phase Cohort 3 (Experimental): Participants who did not achieve clinical response per PCDAI at Week 12 of Period 1 will receive an extended treatment with open-label upadacitinib Dose C daily for an additional 12 weeks. If they are responders after 12 weeks extended treatment, they will continue, otherwise they may be discontinued at the discretion of the investigator
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral Solution/ Extended-Release Tablets
  Other Names: RINVOQ

SUMMARY:
Crohn's disease (CD) is a long-lasting disease that causes severe inflammation (redness, swelling), in the digestive tract, most often affecting the bowels. It can cause many different symptoms including abdominal pain, diarrhea, tiredness, and weight loss. This study will assess how safe and effective oral Upadacitinib is in treating moderately to severely active Crohn's Disease in pediatric participants aged 2 to 18 years old who have had inadequate response, loss of response, intolerance, or medical contraindications to corticosteroids, immunosuppressants, and/or biologic therapy.

Upadacitinib (RINVOQ) is a drug approved in adults for moderate- to severely active CD and is being developed for moderate- to severely active CD in pediatric participants. This study is conducted in 2 periods: Period 1 is comprised of two phases: a 12-week open-label induction phase which means that the study doctor and participants know that participants will receive UPA Dose-A (or the adult equivalent based on body weight) followed by a 52-week double-blind maintenance phase meaning that neither the participants nor the study doctors will know which dose of upadacitinib will be given(UPA Dose B or Dose C). Period 2 is a 156-week open-label extension of Period 1. Approximately 110 pediatric participants with moderate to severely active CD will be enrolled at approximately 92 sites worldwide.

Participants will receive upadacitinib oral tablets once daily or oral solution twice daily at approximately the same time each day, with or without food. Participants will have a safety follow up for 30 days after discontinuation from any time point within the study.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular (weekly, monthly) visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Weight at Screening and Baseline must be ≥ 10 kg
* Moderate to severe CD defined as PCDAI > 30 and endoscopic evidence of mucosal inflammation as documented by a centrally read SES-CD of >/ 6 (or SES-CD of >/4 for isolated ileal disease) excluding the presence of narrowing component.
* Documented diagnosis of CD prior to Baseline, confirmed by colonoscopy during the screening period, with exclusion of current infection, colonic dysplasia and/or malignancy. Appropriate documentation of biopsy results consistent with the diagnosis of CD, in the assessment of the investigator, must be available
* Demonstrated an inadequate response, loss of response, or intolerance to corticosteroids, IMMs, and/or biologic therapy or in whom use of those therapies is medically contraindicated. For participants in the US and South Korea, participants must have demonstrated an inadequate response, loss of response, or intolerance to one or more anti-TNFs (tumor necrosis factor).

Exclusion Criteria:

* History of:

  * A diagnosis of CD prior to 2 years of age.
  * Currently known complications of CD such as:
  * Active abscess (abdominal or perianal);
  * Symptomatic bowel strictures;
  * More than 2 missing segments of the following 5 intestinal segments: terminal ileum, right colon, transverse colon, sigmoid and left colon, and rectum;
  * Ostomy or ileoanal pouch;
  * Surgical bowel resection within the past 3 months prior to Baseline, or a history of more than 3 bowel resections.
* Japan participants only: positive result of beta-D-glucan or two consecutive indeterminate results of beta-D-glucan during the Screening period (screening for Pneumocystis jiroveci infection)
* History of any of the following:

  * Current diagnosis of UC, indeterminate colitis, or monogenic IBD;
  * Fulminant colitis or toxic megacolon;
  * Gastrointestinal perforation (other than due to appendicitis or mechanical injury), diverticulitis, or significantly increased risk for GI perforation per investigator judgment including history of volvulus and/or intussusception (telescoping of bowels);
* Current diagnosis of any primary immune deficiency
* Conditions that could interfere with drug absorption including but not limited to short bowel syndrome or gastric bypass surgery; subjects with a history of gastric banding/segmentation are not excluded.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieved clinical response per the Pediatric Crohn's Disease Activity Index (PCDAI) at Week 12, with clinical remission per the PCDAI at Week 64 | At Week 64
  PCDAI is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Achievement of endoscopic response at Week 64 in participants who achieved clinical response per PCDAI at Week 12. | At Week 64
  Endoscopic response is defined as > 50% reduction in Simple Endoscopic Score for Crohn's Disease (SES-CD) score from Baseline (or for participants with a Baseline SES-CD of 4, at least a 2-point reduction from Baseline), as scored by a central reader.
Number of Participants with Adverse Events | Through Week 156
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related.

SECONDARY OUTCOMES:
Achievement of clinical remission per PCDAI | Week 12
  Clinical remission per PCDAI is defined as PCDAI ≤ 10.
Achievement of endoscopic response | Week 12
  Endoscopic response is defined as > 50% reduction in SES-CD score from Baseline (or for participants with a Baseline SES-CD of 4, at least a 2-point reduction from Baseline), as scored by a central reader.
Achievement of endoscopic remission | Week 12
  Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no subscore > 1, as scored by a central reader
Achievement of clinical response per PCDAI | Week 12
  Clinical response is defined as reduction in PCDAI of ≥ 15 points from Baseline
Achievement of clinical response per PCDAI at Week 64 in participants who achieved clinical response per PCDAI at Week 12 | Week 64
Achievement of endoscopic remission at Week 64 in participants who achieved clinical response per PCDAI at Week 12 | Week 64
  Endoscopic remission is defined as SES-CD ≤ 4 with at least a 2-point reduction from Baseline and no subscore > 1, as scored by a central reader
Achievement of corticosteroid (CS)-free clinical remission per PCDAI at Week 64 in participants who achieved clinical response per PCDAI at Week 12 | Week 64
  CS-free clinical remission per PCDAI: clinical remission per PCDAI and not receiving corticosteroids at Week 12 (for Period 1 induction endpoint[s]); or for at least 90 days prior to the study visit at which endpoint is assessed (for Period 1 maintenance endpoint[s] and Period 2 endpoint[s]).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (83):
- United States (12):
  - UCSF Benioff Children's Hospital - Oakland /ID# 262217, Oakland, California
  - Lucile Packard Children's Hospital /ID# 262193, Palo Alto, California
  - Children's Hospital Colorado - Aurora /ID# 262207, Aurora, Colorado
  - Connecticut Children's Medical Center - Hartford /ID# 262256, Hartford, Connecticut
  - OSF St. Francis Medical Center /ID# 262192, Peoria, Illinois
  - Indiana University Health Riley Hospital for Children /ID# 262215, Indianapolis, Indiana
  - Boston Children's Hospital /ID# 262191, Boston, Massachusetts
  - MNGI Digestive Health, P. A. /ID# 262204, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai /ID# 262216, New York, New York
  - Univ NC Chapel Hill /ID# 262198, Chapel Hill, North Carolina
  - UH Cleveland Medical Center /ID# 262188, Cleveland, Ohio
  - Children's Hospital of Philadelphia - Main /ID# 262197, Philadelphia, Pennsylvania
- Australia (5):
  - Sydney Children's Hospital /ID# 262352, Randwick, New South Wales
  - Children's Hospital at Westmead /ID# 262350, Westmead, New South Wales
  - Queensland Children's Hospital /ID# 262351, South Brisbane, Queensland
  - Monash Health - Monash Medical Centre /ID# 262878, Clayton, Victoria
  - Perth Children'S Hospital /ID# 272905, Perth, Western Australia
- Belgium (6):
  - Uza /Id# 261745, Edegem, Antwerpen
  - Cliniques Universitaires UCL Saint-Luc /ID# 261741, Brussels, Brussels Capital
  - Universitair Ziekenhuis Leuven /ID# 261740, Leuven, Vlaams-Brabant
  - Hospital Universite Enfants Reine Fabiola /ID# 261744, Brussels
  - CHR de la Citadelle /ID# 261749, Liège
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 261750, Namur
- Brazil (5):
  - Galileo Medical Research Ltda /ID# 262602, Juiz de Fora, Minas Gerais
  - Hospital Pequeno Príncipe /ID# 262600, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre /ID# 262601, Porto Alegre, Rio Grande do Sul
  - Rocco & Nazato Servicos Medicos /ID# 262485, São Paulo, São Paulo
  - Hospital Sirio Libanes /ID# 262670, São Paulo
- Bulgaria (2):
  - UMHAT Sveti Georgi /ID# 262590, Plovdiv
  - Specialized Hospital For Active Treatment Of Children Diseases Prof. Ivan Mitev /ID# 262589, Sofia
- IWK Health Center /ID# 262543, Halifax, Nova Scotia, Canada
- China (10):
  - Beijing Children's Hospital /ID# 262258, Beijing, Beijing Municipality
  - Guangzhou Medical University Affiliated Women and Children's Medical Center /ID# 262596, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 272807, Guangzhou, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital /ID# 262300, Zhengzhou, Henan
  - Hunan Children's Hospital /ID# 262512, Changsha, Hunan
  - Jiangxi Provincial Children's Hospital /ID# 262295, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University /ID# 262301, Shenyang, Liaoning
  - Children's Hospital of Shanghai /ID# 262356, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 262502, Shanghai, Shanghai Municipality
  - The Children's Hospital of Zhejiang University School of Medicine /ID# 262337, Hangzhou, Zhejiang
- France (3):
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 262311, Caen, Calvados
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant /ID# 263422, Bron, Rhone
  - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - CHU /ID# 262308, Paris
- Greece (3):
  - Agia Sofia Hospital /ID# 261792, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 261790, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 261791, Heraklion, Crete
- Italy (4):
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 262384, San Giovanni Rotondo, Foggia
  - Ospedale Pediatrico Bambino Gesù /ID# 262379, Rome, Roma
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 262380, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 275276, Milan
- Japan (10):
  - Tsujinaka Hospital - Kashiwanoha /ID# 262454, Kashiwa-shi, Chiba
  - Kurume University Hospital /ID# 262455, Kurume-shi, Fukuoka
  - Miyagi Children's Hospital /ID# 262459, Sendai, Miyagi
  - Osaka Women's and Children's Hospital /ID# 262549, Izumi-Shi, Osaka
  - Saga University Hospital /ID# 262753, Saga, Saga-ken
  - Saitama Children's Medical Center /ID# 262461, Saitama-shi, Saitama
  - Institute of Science Tokyo Hospital /ID# 262510, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Children's Medical Center /ID# 262550, Fuchu-shi, Tokyo
  - National Center For Child Health And Development /ID# 262456, Setagaya City, Tokyo
  - Toyama Prefectural Central Hospital /ID# 262739, Toyama, Toyama
- New Zealand (2):
  - Christchurch Hospital. /ID# 262577, Christchurch, Canterbury
  - Starship Child Health /ID# 262576, Auckland
- Poland (2):
  - Gastromed Sp. z o.o /ID# 262367, Torun, Kuyavian-Pomeranian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 262366, Warsaw, Masovian Voivodeship
- Puerto Rico (3):
  - Clinical Research Investigator Group, LLC /ID# 262357, Bayamón
  - Puerto Rico Health Institute /ID# 262358, Dorado
  - Clinical Research Puerto Rico /ID# 279595, San Juan
- South Korea (3):
  - Seoul National University Hospital /ID# 262324, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 262721, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 262323, Seoul, Seoul Teugbyeolsi
- Spain (5):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 262226, Ferrol, A Coruna
  - Hospital Sant Joan de Deu /ID# 262599, Esplugues de Llobregat, Barcelona
  - Hospital Regional Universitario de Malaga /ID# 262228, Málaga
  - Hospital Universitario Virgen del Rocio /ID# 262712, Seville
  - Hospital Clinico Universitario Lozano Blesa /ID# 262227, Zaragoza
- Taiwan (2):
  - National Taiwan University Hospital /ID# 261695, Taipei City, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 261696, Taoyuan
- United Kingdom (5):
  - Addenbrookes Hospital /ID# 262707, Cambridge, Cambridgeshire
  - Sheffield Children's Hospital NHS Foundation Trust /ID# 261832, Sheffield, England
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 262811, London, Greater London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 262778, Norwich, Norfolk
  - Royal Hospital for Children and Young People /ID# 262388, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M14-671